CLINICAL TRIAL: NCT03287635
Title: Study Title: A Phase 4 Study to Assess the Clinical Efficacy of H.P. Acthar Gel 80 U/ml to Improve the Signs and Symptoms in Subjects With Dry Eye Disease
Brief Title: Clinical Efficacy of H.P. Acthar Gel 80 U/ml to Improve the Signs and Symptoms in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Toyos Clinic (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMT-4223
Record Dates: First submitted 2017-08-28; First posted 2017-09-19 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acthar gel 80 U/ml (Experimental): Patients who continue to experience clinically significant symptoms of dry eye disease even after utilizing traditional methods of treatment for dry eye including but not limited to artificial tears, warm compresses, topical anti-inflammatories like cyclosporine and/or lifitegrast. Patients will receive repository corticotropin intramuscular injections 80 u/ml 2-3 times weekly for up to 3 months as judged by the investigator.
  Interventions: Drug: Corticotropin 80Unit/Ml Repository Injection

INTERVENTIONS:
Drug: Corticotropin 80Unit/Ml Repository Injection — H.P. Acthar Gel (repository corticotropin injection) is an adrenocorticotropic hormone (ACTH) analogue used for: Treatment during an exacerbation or as maintenance therapy in selected cases of systemic lupus erythematosus.
  Other Names: H.P. Acthar gel

SUMMARY:
Study Title: A Phase 4 Study to Assess the Clinical Efficacy of H.P. Acthar Gel 80 U/ml to Improve the Signs and Symptoms in Subjects with Dry Eye Disease

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to investigate the safety and efficacy of H.P. Acthar Gel 80 U/ml in subjects with a documented clinical diagnosis of dry eye disease.

Study Population: The study population will consist of subjects diagnosed with dry eye disease.

Number of Subjects: Approximately 12 subjects

Investigational Product: H.P. Acthar Gel 80 U/ml sufficient for the duration of the study will be supplied by Mallinkrodt to the enrolled subjects

Route and Duration of Administration: Product will be injected subcutaneously weekly by subjects for approximately 12 weeks.

Study Design: This is a Phase 4, single center single arm study designed to evaluate the safety and efficacy of H.P. Achthar Gel in subjects with dry eye disease.

Approximately 25 subjects will be screened and 12 subjects enrolled at one center in the United States.

Subjects will be given 80 international units of study medication subcutaneously depending on the severity of the disease as determined by the primary investigator.

The study will include 3 study visits over 12 weeks. At Visit 1 Screening (14 +/- 1 days prior to Day 1), subjects meeting inclusion/exclusion criteria will begin investigational drug use. Subjects will return for evaluations at Visit 2 (Day 42+/-3 days) and Visit 3 (Day 84 +/-5 days). Subjects will be released from the study at the end of Visit 3 (Day 84+/- 5 days.)

ELIGIBILITY:
Inclusion Criteria:

* At Visit 1 (Screening) individuals of either gender or race will be eligible for study participation if they

  1. Provide written informed consent and HIPAA authorization prior to any study related procedures
  2. Are 18 years of age or older
  3. Are willing and able to follow instructions and can be present for required study visits.
  4. Have documented clinical diagnosis of dry eye disease in one or both eyes.
  5. Have a score of at least 40mm on the ocular discomfort scale
  6. Have at least 5 spk on one or both corneas
  7. Have a grade of 1 or greater in the nasal or temporal areas of one or both eyes.
  8. Have normal lid anatomy.
  9. Are women of child bearing potential who are not pregnant or lactating and who are either abstinent and willing to remain so for the course of the trial or have an IUD in place for at least 3 months prior and through Visit 4, barrier method with spermicide for at least 3 months prior and through Visit 4, stable hormonal contraceptive for at least 3 months prior and through Visit 4 or in a monogamous relationship with a surgically sterilized (vasectomized) partner at least 6 months prior to Visit 1 and through the course of the trial.
  10. Are postmenopausal (no menstrual cycle for at least one year prior to Visit 1) or have undergone bilateral tubal ligation, hysterectomy, hysterectomy with uni or bilateral oophorectomy, or bilateral oophorectomy.

      Exclusion Criteria:

      In order for subjects to be eligible for the study

  <!-- -->

  1. Have a known hypersensitivity or contraindication to the investigational product or their components.
  2. Have used any of the following medications within 14 days prior to screening

     a. Topical or nasal vasoconstrictors
  3. Subjects can be on the following medications if they have been on a stable dose for 12 weeks topical cyclosporine, topical lifitegrast and/or topical loteprednol etabonate. Tetracycline compounds, omega 3s, anticholinergics, anticonvulsants, antidepressants, retinoids, systemic immunosuppressive agents including oral corticosteroids, non-steroidals, antihistamines or mast cell stabilizers, punctal plugs, contact lens wear and glaucoma medications.
  4. Subjects must be unwilling to abstain from eyelash growth medications for the duration of the trial.
  5. Subjects must not have had penetrating intraocular surgery, refractive surgery or corneal transplantation, eyelid surgery within 12 weeks prior to Visit 1.
  6. Subjects with a history of herpetic keratitis.
  7. Have serious or severe disease or uncontrolled medical condition that in the judgement of the investigator could confound study assessments or limit compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Toyos, MD, Principal Investigator — Toyos Clinic
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Toyos M, Toyos R, Jodoin B, Bunch R. Results from a Prospective, Open-Label, Phase 4 Pilot Study of Repository Corticotropin Injection for Moderate and Severe Dry Eye Disease. Ophthalmol Ther. 2022 Jun;11(3):1231-1240. doi: 10.1007/s40123-022-00501-2. Epub 2022 Apr 23. PMID 35460497

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional subjects were added when study participants dropped out due to subject withdrawal, were lost to follow up and physician decision.
Period: Overall Study
Arm/Group | Acthar Gel 80 U/ml
Started | 19
Completed | 12
Not Completed | 7
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Patients experience persistent symptomatic dry eye disease despite treatment with traditional therapies.
Arm/Group | Acthar Gel 80 U/ml
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 54 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Dry Eye Comfort Questionnaire, SANDE
Description: Subjects will be asked to subjectively rate their eye dryness at Visit 1,2 and 3. Subjects will be instructed to rate eye dryness using the scale below. The total length of the line from "no dryness" to "maximal dryness" is 100 mm. The length of the line between the "no dryness" starting point and the first point at which the subject mark crosses the line will be measured in mm. This assessment is a general assessment of the change of both eyes of dryness measure from baseline to final study visit. The measure of discomfort was for the instantaneous measurement at the time of the specific visit.
Time Frame: 12 weeks total. Measure is change on SANDE scale (0 is no dryness and 100mm is maximal dryness) from baseline to final value. Higher values reflect greater amounts of subjective dryness.
Population: Patients receiving Acthar gel injections for 90 days were analyzed
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Acthar Gel 80 U/ml
Number analyzed (Participants) | 12
scores on a scale | 44.77 (3.13)

2. Primary Outcome: 1. Conjunctival Staining With Lissamine Green
Description: Change in Conjunctival staining with lissamine green.
Time Frame: 12 weeks total. Measure is change from baseline to final,
Population: Patients who received Acthar gel SC for 90 days
Measure: Mean (Standard Deviation); unit: staining spots on conjunctiva
Arm/Group | Acthar Gel 80 U/ml
Number analyzed (Participants) | 12
staining spots on conjunctiva | -173.33 (464.59)

3. Secondary Outcome: Intraocular Pressure
Description: goldmann tonometry used by qualified technician with fluorescein staining
Time Frame: 12 weeks measuring change from baseline to final
Population: Patients who received Acthar gel SC or IM for 90 days.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Acthar Gel 80 U/ml
Number analyzed (Participants) | 12
mm Hg | -1.65 (1.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Acthar Gel 80 U/ml
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar Gel 80 U/ml (N=19)
hypertension (Cardiac disorders) | 1 (1) — patient withdrew due to elevated blood pressure. PI unclear if drug related, PI and study participant agreed to stop trial as a precaution and follow for safety. No further events.

LIMITATIONS AND CAVEATS:
single site, open label study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03287635/Prot_004.pdf
  • Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03287635/SAP_005.pdf
  • Informed Consent Form (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT03287635/ICF_006.pdf